CLINICAL TRIAL: NCT04850222
Title: Can Fluoxetine Mitigate the Mental Health Decline Seen in Patients With Musculoskeletal Trauma?
Brief Title: Fluoxetine Mitigation Mental Health Study for Patients With Musculoskeletal Trauma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB202100808; OCR40926 (Other: UF OnCore)
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Musculoskeletal Injury
MeSH Terms: interventions — Fluoxetine; Calcium

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Researchers collecting survey data will be blinded to patients' intervention status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Subjects randomized to get Fluoxetine therapy (Experimental): Subjects will be randomized to take Fluoxetine (10mg by mouth per day). The randomized drug will be prescribed by the orthopedic team on the day randomization so that the patient may be monitored for side effects during the remainder of their hospitalization. The patient will be prescribed the randomized medication on the day of discharge and a 90 day supply will be provided by the inpatient research pharmacy.
  Interventions: Drug: Fluoxetine
- Subjects randomized to get Calcium Supplmentation (Active Comparator): Subjects will be randomized to take Calcium supplementation (1000mg by mouth per day). The randomized drug will be prescribed by the orthopedic team on the day randomization so that the patient may be monitored for side effects during the remainder of their hospitalization. The patient will be prescribed the randomized medication on the day of discharge and a 90 day supply will be provided by the inpatient research pharmacy.
  Interventions: Drug: Calcium

INTERVENTIONS:
Drug: Fluoxetine — Subjects will be randomized to take Fluoxetine (10mg by mouth per day). The randomized drug will be prescribed by the orthopedic team on the day randomization so that the patient may be monitored for side effects during the remainder of their hospitalization. The patient will be prescribed the randomized medication on the day of discharge and a 90 day supply will be provided by the inpatient research pharmacy.
  Arms: Subjects randomized to get Fluoxetine therapy
Drug: Calcium — Subjects will be randomized to take Calcium supplementation (1000mg by mouth per day). The randomized drug will be prescribed by the orthopedic team on the day randomization so that the patient may be monitored for side effects during the remainder of their hospitalization. The patient will be prescribed the randomized medication on the day of discharge and a 90 day supply will be provided by the inpatient research pharmacy.
  Arms: Subjects randomized to get Calcium Supplmentation

SUMMARY:
Musculoskeletal trauma is one of the leading causes of disability in the United States and its negative quality of life impact extends beyond that of physical recovery. More than 50% of victims of musculoskeletal trauma suffer lasting mental health issues following their injury. These symptoms can develop across all spectrums of patients with a variety of injury severities. Previously, this research team developed a ten-step program with the aim of developing fostering coping mechanisms in trauma patients. We were unable to demonstrate a measurable benefit to their mental health or physical function. This has been mirrored in other studies as well; talk therapy and support groups are not a strong enough intervention for some patients.

We hypothesize that a subset of the trauma population would benefit from medical treatment for their depressive and anxious symptoms in the early recovery period. Given the limited resources of mental health systems, it would be ideal for their surgical providers to be able to manage safely their post-injury mental health issues during their surgical follow up. This is a pragmatic pilot study to develop an effective, acceptable, time-limited treatment strategy that could be safely implemented by non-mental health care providers for victims of musculoskeletal trauma.

DETAILED DESCRIPTION:
Rationale

Over 50% of victims of musculoskeletal trauma suffer prolonged depressive and anxious symptomology following their initial injury. This is an independent risk factor for prolonged mental and physical disability. In previous research by the study team in orthopedic trauma patients without previous diagnosis of psychiatric illness, we have demonstrated 28% of these patients had depressive symptomology and 40% had anxiety symptomology 3 months following their traumatic injury. [1] Mental health resources are limited, placing the bulk of patient care on the orthopedic surgeons and primary care physicians. Support groups, self-help programs and talk therapy, while valuable, have not demonstrated measurable efficacy for this patient population. We hypothesize that a subset of the trauma population would benefit from medical treatment for their depressive and anxious symptoms in the early recovery period.

Specific Aims

Aim 1: Evaluate the efficacy of immediate Fluoxetine therapy versus standard of care Calcium treatment in improving mental health and wellbeing in the post-injury period for patients with musculoskeletal trauma.

Hypothesis: Patients randomized to Fluoxetine will have less severe depression, anxiety and post-traumatic stress symptoms than those treated with calcium.

Methodology: Patients >18 years of age admitted to UF Health with extremity fracture(s) resulting from high energy trauma (more than ground level fall) will be enrolled during their index hospitalization. Baseline mental well-being surveys will be obtained (Table 1) and patients will be randomized to calcium supplementation or Fluoxetine. The medications will be started during the hospitalization and prescribed upon discharge. The patient will be followed in the orthopedic clinic on a standard of care post-operative schedule (2 weeks, 3 months, 6 months, and 12 months). Serial mental well-being surveys will be administered at these time points. Post-operative complications such as infection, nonunion or any other reason for return to the operating room will be tracked.

Aim 2: Develop a safe Fluoxetine treatment protocol with a goal to be therapeutic by 6 weeks and taper completely off of treatment by 6-12 months.

Hypothesis: We will be able to develop a standardized, time-limited protocol that could feasibly be utilized by non-mental health providers.

Methodology: Dr. Barbosa De Faria will monitor symptoms and side effects of the Fluoxetine treatment study arm. Any evidence of escalation of depressive or suicidal ideology in either study population will result in immediate psychiatric treatment. Common side effects, medication adherence and appropriate discontinuation will be tracked. Patient reported pain scales will be obtained at each clinic visit as well as documentation of narcotic and cannabis pain treatment during recovery. Patients will be informed of the finite nature of the medical management. We will assess how many patients in the Fluoxetine arm report worsening of symptomology after the cessation of therapy at 9 months and how many seek continued management.

ELIGIBILITY:
Inclusion Criteria:

* patients 18 and older under the care of the UF Orthopedic Trauma Division admitted to UF Health for trauma resulting in one or more extremity or pelvic fractures requiring surgery will be screened.

Exclusion Criteria:

* patients with Traumatic Brain Injury or a past medical history of bipolar or other mental health conditions on current medical management will be excluded
* patients unlikely to follow up (live in at a distance from Gainesville, incarcerated etc.) will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 73 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Serial mental well-being surveys in the post-injury period for patients with musculoskeletal trauma. | Baseline up to 12 months

SECONDARY OUTCOMES:
Patient reported pain scores (PEG score) will be recorded at each visit. | Baseline up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hagen, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lossada-Soto E, Pazik M, Horodyski MB, Vasilopoulos T, de Faria LB, Mathews C, Hagen J. Can fluoxetine mitigate mental health decline in musculoskeletal trauma patients: a pilot single-center randomized clinical trial. Pilot Feasibility Stud. 2022 Aug 17;8(1):184. doi: 10.1186/s40814-022-01119-8. PMID 35978446